CLINICAL TRIAL: NCT03567837
Title: Fructose-induced Hepatic De Novo Lipogenesis in Adolescents With Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was stopped due to the inability to recruit during the Covid epidemic.
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other); University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 180401921
Record Dates: First submitted 2018-06-11; First posted 2018-06-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Fructose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese Metabolically Healthy (Active Comparator): Intervention: Oral challenge of Fructose+Glucose Beverage 1:1, 3g/kg
  Interventions: Other: Fructose + Glucose Beverage
- Obese Pre-diabetes (Experimental): Intervention: Oral challenge of Fructose+Glucose Beverage 1:1, 3g/kg
  Interventions: Other: Fructose + Glucose Beverage

INTERVENTIONS:
Other: Fructose + Glucose Beverage — The intervention is an oral sugar challenge with blood sampling over three hours.

SUMMARY:
In the U.S., dietary fructose has increased in parallel with the increase in obesity and may promote the development of diabetes and other chronic diseases. The largest source of dietary fructose is sweetened beverages that are consumed by adolescents more than any other age group.

This protocol will compare the rates of hepatic de novo lipogenesis (DNL), a process in the liver that changes sugar into fat, in two groups of obese adolescents - one with prediabetes and the other, metabolically healthy. Blood will be sampled before and hourly for 3 hours after the consumption of a fructose-containing beverage. We hypothesize that the pre-diabetic group will show greater DNL in response to fructose. This would support other evidence that increased fructose-induced hepatic DNL is an early mechanism linking dietary sugar to the adverse metabolic sequelae of obesity, including diabetes, fatty liver, dyslipidemia and coronary disease.

DETAILED DESCRIPTION:
Hypothesis: Hepatic DNL in response to the ingestion of fructose:glucose 1:1 is significantly greater in adolescents with obesity and prediabetes compared to adolescents with obesity who are metabolically healthy.

Thirty obese adolescents, ages 12-21 years, will be recruited to each of two groups: 1) prediabetes (n=15) and 2) metabolically healthy (n=15). An attempt will be made to achieve similar age, sex and BMI distributions in the two groups.

Visit 1- Screening: Eligible subjects will be enrolled after Informed consent/assent are obtained by a physician investigator. The medical history will be reviewed and a physical exam performed, including an assessment of pubertal status. Blood will be sampled after at least a 12 hour fast (except water) for complete blood count, serum glutamate pyruvate, glucose, HbA1C, and lipid panel, if not previously documented in the medical record within three months of the screening visit. These tests may be done without fasting, but if the glucose or lipid results are not normal, these two tests must be repeated after fasting.

Visit 2 - Sugar Challenge Test with Blood Sampling: Within three months of the screening visit, eligible participants will return after at least a 12 hour fast (except water). General health, family history and recent diet will be reviewed. The height, weight, waist circumference at the umbilicus, and blood pressure will be recorded. A urine sample will be obtained for microalbuminuria. After placement of an intravenous catheter and withdrawal of the baseline blood samples, participants will drink a sweet beverage prepared by a dietician (fructose:glucose 1:1, 3g/kg, in water). Blood sampling will continue every hour for three hours( ~12 mL per time point).

Percent body fat will be measured by bioimpedance. The percent body fat will be calculated by computer software with prediction equations validated in the pediatric and adult age ranges.

Plasma samples will be obtained at 4 time points (0, 1, 2 and 3 hours), the fatty acid composition of plasma very low density lipoprotein triglyceride (VLDL TG), including %palmitate (16:0), will be measured. A lipid panel and VLDL triglycerides and apolipoprotein B levels will also be measured at each time point. Other assays to be performed include insulin and and glucose, HbA1C and high sensitivity C reactive protein (hsCRP, a marker of inflammation). The urine sample will be assayed for microalbuminuria (albumin/creatinine >30 mg/g).

An interim analysis of the primary endpoint (increase in VLDL TG %16:0) will be performed in the first three subjects of each group to determine whether the dose of sugar and sampling duration of 3 hours are sufficient to produce a measurable increase in VLDL TG %16:0.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 12-21 years old.
2. BMI percentile >95th and <140th percentile of the 95th, maximum weight 110 kg.
3. Group 1: HbA1C <5.7% and no history of fasting hyperglycemia (glucose greater or equal to100 mg/dL and/or HbA1C greater or equal to 5.7%), sustained hypertension (>95th percentile) or abnormal lipids (LDL cholesterol <130 mg/dL, TG <130 mg/dL, HDL-C >40 mg/dL).

   Group 2: HbA1C greater or equal to 5.7 to 6.49%
4. Pubertal or post- pubertal stage (pre-pubertal excluded).
5. Willing and able to stop fish oil, fiber supplement, other non-prescribed vitamins/supplements for 1 week prior to study visit.
6. Willing to not drink alcohol for at least 48 hours before the study visit.
7. Willing to refrain from vigorous exercise the day before the study visit.

Exclusion Criteria:

1. Diabetes (fasting blood glucose greater or equal to126 mg/dL, and/or HbA1C >6.5% and/or history of a 2 hour oral glucose tolerance test (OGTT) >200 mg/dL).
2. Triglycerides >500 mg/dL, LDL cholesterol >160 mg/dL.
3. Medications affecting lipid or glucose metabolism, including hormonal contraceptives.
4. Liver disease or intestinal dysfunction. Serum glutamate oxaloacetate and/or serum glutamate pyruvate < 2x upper limit normal is permitted if there is no diagnosis of liver disease by a gastroenterologist.
5. Weight loss >10% in past 6 months.
6. Cigarette smoking.
7. Alcohol or drug abuse.
8. Systemic illness, including polycystic ovary disease and acute infections within two weeks of study visits.
9. Anemia.
10. Pregnancy or breast feeding.
11. Psychiatric illness.
12. Extreme diet or level of physical activity.
13. Fructose intolerance.
14. Implanted electronic devices (bioimpedance measurement).
15. Any other condition, which in the opinion of the principal investigator, should prohibit participation in the study.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Increase in VLDL TG palmitate | Three hours
  In the 2 study groups: a comparison of the increase in VLDL TG palmitate over 3 hours after ingestion of a beverage made with fructose and glucose.
  after an oral challenge of fructose+glucose

SECONDARY OUTCOMES:
Correlation of the increase in VLDL TG palmitate and markers of carbohydrate and fatty acid metabolism | Three hours
  In the two study groups: a comparison of other markers of carbohydrate and fatty acid metabolism (i.e. VLDL and total TG, cholesterol, apolipoprotein B, insulin, and glucose) before and after the oral sugar challenge.
  2) To correlate these markers with the increase in VLDL TG %16:0.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hudgins, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- Weill Cornell Medicial College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No